CLINICAL TRIAL: NCT05048199
Title: Hemodynamic Effects of Pressure-regulated Volume Controlled Versus Volume-controlled Ventilation Mode in Patients With Diastolic Dysfunction Undergoing Radical Cystectomy- A Cross Over Randomized Study
Brief Title: Hemodynamic Effects of Pressure-regulated Volume Control Mode in Patients With Diastolic Dysfunction Undergoing Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mahmoud Othman, Professor of anesthesia and surgical Intensive care, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: MD.21.07.479.R1
Record Dates: First submitted 2021-08-26; First posted 2021-09-17 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Radical Cystectomy
Keywords: Diastolic dysfunction; Pressure regulated volume control mode; Cardiac output

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pressure regulated volume-controlled mode of ventilation (PRVC group) (Experimental): The mode selected for mechanical ventilation is settled by randomization either PRVC or VCV during radical cystectomy, then the mode of ventilation will be switched to the other mode during urinary diversion till the end of surgery according to the randomization sequence. The tidal volume in both groups will be set to deliver 6-8 mL/kg of ideal body weight. The respiratory rate (RR) will be adjusted to maintain an end tidal CO2 (ETCO2) level of 30-35 mmHg, the inspiratory to expiratory time (I: E) ratio will be1:2 and PEEP 5-8 cmH2O.
  Interventions: Device: pressure regulated volume-controlled mode of ventilation
- volume-controlled mode of ventilation (VC group) (Active Comparator): The mode selected for mechanical ventilation is settled by randomization either PRVC or VCV during radical cystectomy, then the mode of ventilation will be switched to the other mode during urinary diversion till the end of surgery according to the randomization sequence. The tidal volume in both groups will be set to deliver 6-8 mL/kg of ideal body weight. The respiratory rate (RR) will be adjusted to maintain an end tidal CO2 (ETCO2) level of 30-35 mmHg, the inspiratory to expiratory time (I: E) ratio will be1:2 and PEEP 5-8 cmH2O.
  Interventions: Device: volume-controlled mode of ventilation

INTERVENTIONS:
Device: pressure regulated volume-controlled mode of ventilation — Cardiac output non-invasive monitor for measuring SV. Hemodynamic variables including heart rate (HR), mean arterial blood pressure (MAP), central venous pressure (CVP), stroke volume (SV), stroke volume index (SVI), cardiac output (COP), cardiac index (CI), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI), thoracic fluid content (TFC), corrected flow time (FTC), index of contractility (ICON), and systolic time ratio (STR), Arterial oxygen saturation (Sao2), oxygen delivery (DO2) and oxygen delivery index (DO2I) will be recorded.
  These variables will be obtained before induction of anaesthesia (T1) skin incision (T2), then every 30 min till the resection of the urinary bladder (T3a, T3b, T3c, …. etc). The mode of ventilation will swift to the other mode 5 minutes after cystectomy (T4), then every 30 min till end of the urinary diversion (T5a, T5b, T5c, …. etc), end of surgery (T6), and postoperative every 4h for 24 hours( P1-P6).
  Arms: pressure regulated volume-controlled mode of ventilation (PRVC group)
Device: volume-controlled mode of ventilation — Cardiac output non-invasive monitor will be used for measuring SV. Hemodynamic variables including heart rate (HR), mean arterial blood pressure (MAP), central venous pressure (CVP), stroke volume (SV), stroke volume index (SVI), cardiac output (COP), cardiac index (CI), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI), thoracic fluid content (TFC), corrected flow time (FTC), index of contractility (ICON), and systolic time ratio (STR), Arterial oxygen saturation (Sao2), oxygen delivery (DO2) and oxygen delivery index (DO2I) will be recorded.
  These variables will be obtained before induction of anaesthesia (T1) skin incision (T2), then every 30 min till the resection of the urinary bladder (T3a, T3b, T3c, …. etc). The mode of ventilation will swift to the other mode 5 minutes after cystectomy (T4), then every 30 min till end of the urinary diversion (T5a, T5b, T5c, …. etc), end of surgery (T6), and postoperative every 4 hours for 24 hours (P1-P6).
  Arms: volume-controlled mode of ventilation (VC group)

SUMMARY:
Diastolic function is a combination of ventricular chamber compliance, active myofilament relaxation, and elastic recoil of systolic potential energy. Diastole is classically divided into four stages-isovolumetric relaxation, early rapid filling, late slow filling, and atrial contraction. Isovolumetric relaxation refers to the rapid decrease in LV pressure with little or no change in volume and ends with the opening of the mitral valve and early LV filling. These early phases, sometimes referred to as LV suction, are characterized by a rapid decline in LV intracavity pressure and require energy in the form of ATP to pump cytosolic calcium back into the sarcoplasmic reticulum and enable uncoupling of actin and myosin. Filling later in diastole is more dependent on ventricular compliance.

Up to investigator knowledge, the effect of mechanical ventilation on patient hemodynamics is still unclear especially in patients with diastolic dysfunction. The optimal ventilation mode for anesthesia of patient with diastolic dysfunction remains a subject of debate. The primary outcome of this study is to investigate whether the pressure regulated volume-controlled mode (PRVC) in comparison with the volume-controlled mode in patients with diastolic dysfunction is associated with better hemodynamic alterations and different vasopressors support during anesthesia for radical cystectomy.

DETAILED DESCRIPTION:
Diastolic dysfunction represents an abnormality in left ventricular relaxation and/or compliance that changes the onset, rate and extent of LV pressure decline and filling during diastole. These changes cause an abnormal relation between LV pressure and volume so that higher filling pressures are required to maintain normal LV end-diastolic volume and cardiac output .Ventricular compliance is affected by numerous factors, including the accumulation of cytoskeletal collagen, which increases with age (over 60 years), longstanding wall stress beyond its physiological reserve, for example, during episodes of uncontrolled systemic hypertension, long term DM, obesity, cardiac ischemia or atrial fibrillation (AF), and various neuro-humoral factors. Less common causes are infiltrative diseases, pericardial constriction, and collection. .

Echocardiographic examination of diastolic function including transmitral flow velocities early (E) and atrial (A), as well as the corresponding velocities of the mitral valve annuli (e' and a'), is currently recommended .After cardiac and noncardiac surgery, diastolic dysfunction is thought to be a risk factor for postoperative consequences including greater mortality and a higher incidence of serious cardiovascular events including myocardial infarction, pulmonary edema, ventricular fibrillation, or primary cardiac arrest and complete heart block. However, the underlying mechanism by which diastolic dysfunction raises the risk of postoperative complications is unknown. Anesthetic drugs may cause altered hemodynamic function and subsequent impairment of diastolic function in patients with diastolic dysfunction, which may be linked to a higher incidence of postoperative problems Positive pressure ventilation is required for anesthesia, and significant volume shifts occur intraoperatively and postoperatively, especially in major surgery. The interactions of positive pressure ventilation with the cardiovascular system are complex and affect both ventricles .Whereas Volume-controlled ventilation ensures the delivery of a defined tidal volume and uses a square waveform flow delivery method that produces high peak airway pressures in low-compliance states. On the other hand, Pressure-regulated volume-controlled (PRVC) mode of ventilation is an example of adaptive targeting mode. There is the adaptive targeting of inspiratory pressure with the aim of delivering the desired minute tidal volume. The ventilator uses a feedback method on breath-to-breath basis to continuously adjust the pressure delivered to achieve the tidal volume target .The effects of different ventilatory modes on patient´s hemodynamics requires further investigations, the increase of the intrathoracic pressure produced by mechanical ventilation can decrease venous return and then preload resulting in decreased cardiac output .

Management of hemodynamics remain one of the core tasks in perioperative and critical care settings. The basis of hemodynamic management in patients undergoing major surgery is formed by a rational titration of fluids, vasopressors and inotropes. the use of dynamic parameters to guide intravenous and inotropic therapy is frequently applied with the intention to optimize peri-operative hemodynamic profiles and maximize oxygen delivery in patients undergoing major abdominal surgery .Direct measurement of SV using noninvasive techniques has become an accepted tool for guiding fluid administration in high risk surgical patients. Dynamic indices have emerged as promising predictors in last decade, and have been proven to predict fluid responsiveness far better than static measures .

This prospective, randomized, cross- over study will be conducted on 76 pairs of patients scheduled for radical cystectomy. A written informed consent will be obtained from all participants in the study.This study will include adult patients -who diagnosed by preoperative cardiac ECHO-with diastolic dysfunction of both sexes. The patients at risk of diastolic dysfunction usually include concomitant comorbidities like long term hypertension, diabetes mellitus, atrial fibrillation or aged patients above 65 years who will scheduled for radical cystectomy and urinary diversion for muscle invasive urinary bladder carcinoma at Mansoura Urology and Nephrology Centre (UNC).

ELIGIBILITY:
Inclusion Criteria:

1. adult patients with diagnosed diastolic dysfunction.
2. long term controlled hypertension.
3. Long term controlled diabetes mellitus.
4. Controlled atrial fibrillation.
5. Aged patients above 60 years

Exclusion Criteria:

1. Patients younger than 18 years.
2. Patients with body mass index (BMI) ˂ 25 and ˃35 wts
3. Major cardiovascular problems with ejection fraction ˂ 40 %.
4. Any implanted mechanical cardiac device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
The incidence of noradrenaline use during anesthesia. | perioperative time for 24 hours
  The number of patients that will need noradrenaline as vasopressor during anesthesia with either modes of ventilation to maintain hemodynamic stability.
The incidence of Cardiac output changes during anesthesia . | perioperative time for 24 hours
  The number of participants associated with cardiac output and stroke volume drop during anesthesia with each mode of ventilation .

SECONDARY OUTCOMES:
The incidence of any other inotropic administration during perioperative time | perioperative time for 24 hours
  The number of participants and total dose of other inotropic administration like dobutamine or dopamine during perioperative time to ensure hemodynamic stability.
The incidence of difficult weaning from mechanical ventilation . - | End of surgery.
  The number of participants associated with difficult weaning from mechanical ventilation that may be enhanced by diastolic dysfunction in both groups.
Incidence of associated myocardial ischemia, infarction, arrhythmia or cardiogenic pulmonary edema. | perioperative time for 24 hours.
  Decrease incidence of associated predefined Myocardial ischemia, infarction, arrhythmia, cardiogenic pulmonary edema.
The incidence of postoperative hypotension . | 24-hours postoperative
  The number of participants that will presented with postoperative hypotension with mean arterial blood pressure less than 65 mmHg in both groups
The incidence postoperative mortality. | 7-days postoperative
  The incidence of postoperative mortality of anesthesia related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Othman, Principal Investigator — Department of anesthesia ,Urology and nephrology center ,Faculty of medicine,Mansoura university
Locations (1):
- Urology and nephrology center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No